CLINICAL TRIAL: NCT00375362
Title: The Analgesic Efficacy of Nitroglycerin Patches for Postoperative Pain in Patients Undergoing Total Knee Arthroplasty
Brief Title: The Analgesic Effect of Nitroglycerin Patch for Postoperative Pain After Total Knee Replacement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 004083
Record Dates: First submitted 2006-09-12; First posted 2006-09-13 (Estimated); Last update posted 2006-09-13 (Estimated); Status verified 2006-07

CONDITIONS: Total Knee Arthroplasty
Keywords: nitroglycerin; morphine; patient controlled analgesia; total knee arthroplasty

INTERVENTIONS:
Drug: Nitroderm patch

SUMMARY:
Patients who undergo general anestheesia for total knee arthroplasty pften have sever postoperative pain which hinders their rehabilitation. Nitroglycerin patches have been found to cause alleviation of pain especially when used in conjuction with morphine. Therefore we propose placement of a nitroglycerin patch after total kneee arthroplasty surgery and see how it affects pain scores or causes less nedd for morphine after surgery.

DETAILED DESCRIPTION:
Patients undergoing total knee arthroplasty will be randomized into two groups: control and placebo.

Eache patient will undergo total knee arthroplasty under general anesthesia. Both groups will get the same anesthetic protocal. At the end of surgery, before awakening patients will recieve either a nitroglycerin or placebo patch on their back. Both the participant and the investigator will be blinded to the group assisignment. At the end of surgery both groups will recieve morphine for postoperative pain. In the recovery room they will be given patient controlled analgesia with morphine. An investigator blinded to study assisignment will record pain scores, sedation scores, nauseau and vomiting. Patients will be given patient controlled analgesia for 24 hours and they will be followed for pain levels, morphine use, sedation and nauseau levels. The nitroderm or placebo patch will be removed after 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients undergoing total knee arthroplasty

Exclusion Criteria:

* Pshychiatric disorder
* Allergy to nitroglycerin or morphine
* Chronic renal failure
* Migraine headaches
* Hypotension

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2006-07; Study Completion 2006-09

PRIMARY OUTCOMES:
pain scores
morphine use
sedation score
nausea and vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Leonid A Eidelman, MD, Study Director — Rabin Medical Center; Sharon Orbach-Zinger, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petach Tikvah, Israel